CLINICAL TRIAL: NCT06057181
Title: Helix Research Network
Acronym: HRN
Status: Recruiting | Type: Observational
Sponsor: Helix, Inc (Industry)
Collaborators: Medical University of South Carolina (Other); HealthPartners Institute (Other); Memorial Hermann Health System (Other); WellSpan Health (Other); St. Luke's Hospital and Health Network, Pennsylvania (Other); Sanford Health (Other); Renown Health (Other); WakeMed Health and Hospitals (Other); University of Nebraska (Other); Ohio State University (Other); Cone Health (Other); Parkview Health (Other); Rochester Regional Health (Unknown); University Health Network, Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: HRN 001
Record Dates: First submitted 2023-08-18; First posted 2023-09-28 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Genetic Predisposition to Disease; Genetics Disease
MeSH Terms: conditions — Genetic Predisposition to Disease; Genetic Diseases, Inborn | interventions — Exome Sequencing

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Genetic: Exome sequencing — Exome sequencing will be completed on each sample submitted.

SUMMARY:
The Helix Research Network ("HRN") is a network of academic, public, and/or private healthcare organizations that are committed to advancing medical research and improving human health through large-scale genomics research and acceleration of the integration of genomic and other omics data into clinical care.

DETAILED DESCRIPTION:
The network will create a large-scale clinicogenomics dataset, which will support research to discover molecular and genetic determinants of disease risk, disease progression, treatment response, health economic outcomes, social or behavioral determinants of health, targets for therapeutic intervention, risk stratification, clinical implementation, and other clinical indicators of interest. This clinicogenomics dataset will be used to reveal molecular and/or genetic factors that could improve the diagnosis or medical treatment of individual participants and includes a process to share individual results with participants. Participants will also receive annual reports on study outcomes and the impact of HRN, as such information becomes available.

Institutional membership in HRN will consist of Helix and member healthcare systems (herein referred to as "HRN Member Site(s)"). The Helix Research Network is a multi-center research program that will enroll an unlimited number of participants. Participants will be recruited concurrently from HRN Member Sites. In some cases, HRN Member Sites may recruit participants from multiple clinical sites. Participants who meet the enrollment criteria established in this protocol will be enrolled if they or their legally authorized representative(s) provide informed consent in accordance with all applicable regulations and sIRB requirements. Participants will be enrolled until withdrawal from the study or end of the study. Participants may be recruited at any point during the study period, until the recruitment goals established by the protocol are met.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* Willing and able to comply with all aspects of the protocol

Exclusion Criteria:

* History of allogenic bone marrow transplant
* History of allogenic stem cell transplant
* Anything that would place the individual at increased risk or preclude an individual's: 1) full compliance with study requirements; or 2) completion of the study based on the assessment from local consenting and enrolling Investigators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study will recruit the general population from the surrounding areas of the HRN Member Sites. This may include patients within a health system of the Site or community members in the surrounding area of Sites.
Sampling Method: Non-Probability Sample
Enrollment: 2000000 (Estimated)
Dates: Start 2021-09-13 (Actual); Primary Completion 2031-09-13 (Estimated); Study Completion 2036-09-13 (Estimated)

PRIMARY OUTCOMES:
Establish a Research Network | Through study completion, average 10 years
  Establish a research network to support the advancement of biomedical research, improve human health through genomics research, and accelerate integration of genomic and other omics data into clinical care.
Aggregate data | Through study completion, average 10 years
  Aggregate molecular, genomic data, phenotypic and other health-related data in centralized and/or federated databases to be accessed by investigators for approved research purposes.
Re-Contact participants | Through study completion, average 10 years
  Recontact participants for additional data collection, research participation opportunities, and return of results
Genetic biomarker identification | Through study completion, average 10 years
  Identification and characterization of clinical, histological, molecular, and genetic biomarkers that are linked to disease, disease outcomes, or that might be used to improvise disease classification.
Exploration of genetic determinants of disease | Through study completion, average 10 years
  Exploration of the molecular and genetic underpinnings and determinants of disease, including disease risk, disease progression, treatment response, health economic outcomes, social or behavioral determinants of health, targets for therapeutic intervention, risk stratification, and other clinical indicators of interest.
Collection and analysis of Patient Reported Outcomes | Through study completion, average 10 years
  Collection and analysis of Patient Reported Outcomes (e.g. quality of life, physical function, symptom burden) associated with diseases that have a genetic or molecular etiology. Validation of disease-specific instruments to assess the impact of genetic screening.

CONTACTS AND LOCATIONS:
Overall Officials: William Lee, PhD, Principal Investigator — Helix, Inc
Locations (13):
- United States (13):
  - Parkview Health, Fort Wayne, Indiana
  - HealthPartners (myGenetics), Bloomington, Minnesota
  - Nebraska Medicine - University of Nebraska Medical Center (Genetic Insights Project), Omaha, Nebraska
  - Rochester Regional Health, Rochester, New York
  - Cone Health (Gene Connect), Burlington, North Carolina
  - WakeMed (PreciselyYou), Raleigh, North Carolina
  - TriHealth, Cincinnati, Ohio
  - The Ohio State University (Genomic Health), Columbus, Ohio
  - St. Luke's University Health Network (DNAanswers), Bethlehem, Pennsylvania
  - WellSpan Health (The Gene Health Project), York, Pennsylvania
  - Medical University of South Carolina (In Our DNA SC), Charleston, South Carolina
  - Sanford Health (Imagine You), Sioux Falls, South Dakota
  - Memorial Hermann Health System (genoME), Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
As a population health research network, the primary purpose of HRN is to help researchers and clinicians better understand how genetic information may be used to improve the health of individuals and communities. It is possible that participants may receive actionable health information as a result of analysis of their DNA information. This means that the participant's genetic results may be used by their healthcare providers to inform medical decisions. It is also possible that novel discoveries may be generated from the research that could positively impact a participant's healthcare in the future.
Supporting Information: ICF, CSR
Time Frame: Data will be available for the duration of the study.
Access Criteria: An application to the Helix Research Network or a Member Site for Member Site level data.